CLINICAL TRIAL: NCT03556553
Title: Clinical Evaluation of a Self-Adhering Flowable Composite in Class I Cavities
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Dr. Fatma Dilşad Öz, PhD, DDS, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Vertise-Luxa Flow
Record Dates: First submitted 2018-05-24; First posted 2018-06-14 (Actual); Last update posted 2021-09-14 (Actual); Status verified 2021-09

CONDITIONS: Tooth Diseases
Keywords: composite resin; occlusal caries
MeSH Terms: conditions — Tooth Diseases

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vertise Flow (Experimental): Superficial Class I cavities restored with Vertise Flow
  Interventions: Device: Vertise Flow
- LuxaFlow (Experimental): Superficial Class I cavities restored with LuxaFlow
  Interventions: Device: LuxaFlow; Device: Teco Adhesive

INTERVENTIONS:
Device: Vertise Flow — Composite resin
  Other Names: Self-adhering flowable composite
  Arms: Vertise Flow
Device: LuxaFlow — Composite resin
  Other Names: Flowable composite with Teco adhesive system
  Arms: LuxaFlow
Device: Teco Adhesive — Adhesive system
  Arms: LuxaFlow

SUMMARY:
The aim of this study is to evaluate long-term clinical performance of a self-adhering flowable resin composite in comparison with a conventional flowable resin composite used with an etch&rinse adhesive system in minimally invasive class I cavities. Twenty-five patients will receive at least one pair of class I restorations. After class I cavities were prepared they were restored either with a self-adhering flowable resin composite (VertiseFlow/Kerr-VR) or with a flowable resin composite (Luxaflow/DMG-LX) in combination with an etch&rinse adhesive (Teco/DMG) [according to the manufacturers' instructions. Restorations will be evaluated at baseline and yearly according to FDI criteria by two evaluaters. Statistical analysis will be carried out with Pearson Chi-Square test and Cochran Q-test followed by Mc Nemar's.

ELIGIBILITY:
Inclusion Criteria:

* having no medical or behavioral problems preventing then from attending review visits, absence of previously placed restorations,having antagonist teeth

Exclusion Criteria:

* poor gingival health,uncontrolled, rampant caries,bruxism,removable partial dentures, xerostomia

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2011-03-30 (Actual); Primary Completion 2011-06-30 (Actual); Study Completion 2016-06-30 (Actual)

PRIMARY OUTCOMES:
Clinical performances of flowable composite resins | Five years
  Five year results according to FDIcriteria